CLINICAL TRIAL: NCT03639714
Title: An International Phase 1/2 Study of GRT-C901/GRT-R902, a Neoantigen Cancer Vaccine, in Combination With Immune Checkpoint Blockade for Patients With Advanced Solid Tumors
Brief Title: A Study of a Personalized Neoantigen Cancer Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gritstone bio, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO-004
Record Dates: First submitted 2018-08-06; First posted 2018-08-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Non Small Cell Lung Cancer; Colorectal Cancer; Gastroesophageal Adenocarcinoma; Urothelial Carcinoma
Keywords: neoantigen cancer vaccine; personalized neoantigen cancer vaccine; GRT-C901; GRT-R902; immunotherapy; nivolumab; ipilimumab; PD-1; CTLA-4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Carcinoma, Transitional Cell; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): * GRT-C901
  * GRT-R902
  * nivolumab
  * ipilimumab
  Interventions: Biological: GRT-C901; Biological: GRT-R902; Biological: nivolumab; Biological: ipilimumab
- Phase 2 Cohorts (Experimental): * GRT-C901
  * GRT-R902
  * nivolumab
  * ipilimumab
  Interventions: Biological: GRT-C901; Biological: GRT-R902; Biological: nivolumab; Biological: ipilimumab

INTERVENTIONS:
Biological: GRT-C901 — a patient-specific neoantigen cancer vaccine prime
Biological: GRT-R902 — a patient-specific neoantigen cancer vaccine boost
Biological: nivolumab — anti-PD-1 monoclonal antibody
  Other Names: Opdivo
Biological: ipilimumab — anti-CTLA-4 monoclonal antibody
  Other Names: Yervoy

SUMMARY:
The purpose of this study is to evaluate the safety, dose, immunogenicity and early clinical activity of GRT-C901 and GRT-R902, a personalized neoantigen cancer vaccine, in combination with nivolumab and ipilimumab, in patients with metastatic non-small cell lung cancer, microsatellite stable colorectal cancer, gastroesophageal adenocarcinoma, and metastatic urothelial cancer.

DETAILED DESCRIPTION:
Tumors harboring non-synonymous deoxyribonucleic acid (DNA) mutations can present peptides containing these mutations as non-self antigens in the context of HLA on the tumor cell surface. A fraction of mutated peptides result in neoantigens capable of generating T-cell responses that exclusively target tumor cells. Sensitive detection of these mutations allows for the identification of neoantigens unique to each patient's tumor to be included in a personalized cancer vaccine that targets these neoantigens. This vaccine regimen uses two vaccine vectors as a heterologous prime/boost approach (GRT-C901 first followed by GRT-R902) to stimulate an immune response. This study will explore the safety and early clinical activity of this patient-specific immunotherapy intended to induce T-cell responses specific for neoantigens.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated informed consent form prior to initiation of study-specific procedures.
* Patients with the indicated advanced or metastatic solid tumor as follows:

  1. NSCLC who are planned for or have received no more than 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy (note: patients who have received anti-PD-(L)1 monotherapy are eligible)
  2. GEA who are planned for or have received no more than 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy
  3. mUC who are planned for or have received no more than 1 cycle of systemic treatment with cytotoxic, platinum-based chemotherapy
  4. CRC-MSS who are receiving first line systemic therapy or who are planned for or have received no more than 1 cycle of second line systemic therapy including a fluoropyrimidine and oxaliplatin or irinotecan
* 18 years of age or older
* ECOG Performance Status 0 or 1
* Lesion amenable to biopsy
* Measurable disease according to RECIST v1.1
* Have adequate organ function, as measured by laboratory values (criteria listed in protocol)

Exclusion Criteria:

* Tumors with genetic characteristics as follows:

  1. For NSCLC, patients with a known genetic driver alteration in EGFR, ALK, ROS1, RET, or TRK
  2. For CRC and GEA, patients with known MSI-high disease based on institutional standard
  3. For CRC, patients with a known BRAF V600E mutation or patients with peritoneal carcinomatosis and for GEA, patients with peritoneal carcinomatosis as their only evidence of disease
* Patients with known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Known exposure to chimpanzee adenovirus or any history of anaphylaxis in reaction to a vaccination or allergy or hypersensitivity to study drug components
* Bleeding disorder (eg., factor deficiency, coagulopathy) or history of significant bruising or bleeding following IM injections or blood draws

Complete inclusion and exclusion criteria are listed in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | Initiation of study treatment through 100 days post-last dose (up to approximately 27 months)
Objective Response Rate (ORR) in Phase 2 using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 27 months)
Identify the recommended Phase 2 dose (RP2D) of GRT-C901 and GRT-R902 | Up to approximately 6 months

SECONDARY OUTCOMES:
Measure the immune response to neoantigens encoded by GRT-C901 and GRT-R902 | Baseline to end of treatment (up to approximately 12 months)
Objective Response Rate (ORR) in Phase 1 using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 4 years)
Duration of response (DOR) using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 4 years)
Clinical benefit rate (using RECIST v1.1) | Initiation of study treatment until disease progression (up to approximately 4 years)
Progression-free survival (PFS) | Up to approximately 4 years
Overall survival (OS) | Up to approximately 4 years
Percentage of patients for whom vaccine is successfully manufactured and timeframe for vaccine manufacturing | Study enrollment to initiation of study treatment (up to approximately 6 months)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - The University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Palmer CD, Rappaport AR, Davis MJ, Hart MG, Scallan CD, Hong SJ, Gitlin L, Kraemer LD, Kounlavouth S, Yang A, Smith L, Schenk D, Skoberne M, Taquechel K, Marrali M, Jaroslavsky JR, Nganje CN, Maloney E, Zhou R, Navarro-Gomez D, Greene AC, Grotenbreg G, Greer R, Blair W, Cao MD, Chan S, Bae K, Spira AI, Roychowdhury S, Carbone DP, Henick BS, Drake CG, Solomon BJ, Ahn DH, Mahipal A, Maron SB, Johnson B, Rousseau R, Yelensky R, Liao CY, Catenacci DVT, Allen A, Ferguson AR, Jooss K. Individualized, heterologous chimpanzee adenovirus and self-amplifying mRNA neoantigen vaccine for advanced metastatic solid tumors: phase 1 trial interim results. Nat Med. 2022 Aug;28(8):1619-1629. doi: 10.1038/s41591-022-01937-6. Epub 2022 Aug 15. PMID 35970920